CLINICAL TRIAL: NCT04829279
Title: Evaluation of Effectiveness for Connected Network for EMS Comprehensive Technical-support Using Artificial Intelligence (CONNECT-AI) System by Community Intervention: A Prospective Crossover Interventional Study
Brief Title: Evaluation of Effectiveness for Connected Network for EMS Comprehensive Technical-support Using Artificial Intelligence (CONNECT-AI) System by Community Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 4-2021-0217
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Emergency Patient Transported by Ambulance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental): Emergency patient transferred by CONNECT AI system
  Interventions: Other: CONNECT AI system group
- Control (No Intervention): Emergency patient transferred by conventional EMS

INTERVENTIONS:
Other: CONNECT AI system group — A. During the Intervention period, paramedics wear equipment for multi-faceted data acquisition and press the start button of the system.
  B. During the Intervention period, inside the ambulance, a application that implements a function that automatically evaluates the patient's severity, displays a list of optimal transfer hospitals based on this, and shares real-time information of the hospitals, is installed so that paramedics can refer to the work.
  C. ED's medical staff will receive through ER-kiosk pre-hospital patient information collected and analyzed through the CONNECT AI system before arrival.
  Arms: Case

SUMMARY:
This study aims to verify the effectiveness of the connected network for EMS comprehensive technical-support using artificial intelligence (CONNECT-AI) system through demonstration in the local community. The study was designed as a prospective non-random cross-intervention study design in two preselected communities. The subjects of the study are patients transferred to the local emergency department(ED) through an ambulance of a fire department in the selected community. If the storage and transmission of information collected by an ambulance fails or the information of the transferred patient cannot be verified in the transferred ED, it is excluded from the study. In this study, the developed CONNECT-AI system was installed in all emergency vehicles and EDs in two regional cohorts, and the effectiveness was measured by operating an intersection for the same period. The primary outcome is the transfer time spent in the pre-hospital stage, and the secondary outcome is whether the optimal transfer hospital is selected.

ELIGIBILITY:
Inclusion Criteria:

* patients transferred to the local emergency department(ED) through an ambulance of a fire department in the selected community.

Exclusion Criteria:

* If the storage and transmission of information collected by an ambulance fails or the information of the transferred patient cannot be verified in the transferred ED

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15392 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
transfer time spent in the pre-hospital stage | up to 1 month
  Time taken from the time the paramedic arrives at the scene to the transfer hospital

SECONDARY OUTCOMES:
Whether to select the optimal transfer hospital | up to 1 month
  In the case of transfer to another hospital or death without resolving the emergency situation at the initial ED

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Jae Chang, Principal Investigator — Division of Cardiology, Yonsei university college of medicine
Locations (1):
- Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Kim MJ, Kim HC, Kim HY, Sung JM, Chang HJ. A Novel Artificial Intelligence-Enhanced Digital Network for Prehospital Emergency Support: Community Intervention Study. J Med Internet Res. 2025 Jan 23;27:e58177. doi: 10.2196/58177. PMID 39847421